CLINICAL TRIAL: NCT00661505
Title: A Single Arm Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous C.E.R.A. for the Maintenance of Haemoglobin Levels in Haemodialysis Patients With Chronic Renal Anaemia.
Brief Title: A Study of Intravenous Mircera in Hemodialysis Patients With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21096
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C.E.R.A. 120, 200, or 360 mcg (Experimental): Eligible participants were administered Continuous Erythropoietin Receptor Activator (C.E.R.A.) at a dose of 120, 200, or 360 microgram (mcg), intravenously (IV), every 4 weeks i.e. Weeks 4, 8, 12, 16 and 20 but not on Weeks 24 and 28. The initial dose of C.E.R.A.was based on the last dose of the previous Erythropoiesis Stimulating Agent (ESA). The ESA therapy was administered from enrollment to the 4 weeks stability verification period (SVP), weekly, either as epoetin (<8000 IU, 8000-16000 IU, or >16000 IU) or darbepoetin alpha (<40 mcg, 40-80 mcg, or >80 mcg). A telephone follow-up visit took place 4 weeks after the end of C.E.R.A. treatment (Week 28).
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — 120, 200 or 360 micrograms iv every 4 weeks (starting dose)

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of once-monthly administration of intravenous Mircera for the maintenance of hemoglobin levels in hemodialysis patients with chronic renal anemia. Patients will receive 4-weekly intravenous injections of Mircera, at a starting dose of 120, 200 or 360 micrograms. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >= 18 years of age;
* chronic renal anemia;
* continuous stable iv or sc maintenance epoetin therapy during previous 4 weeks;
* regular long-term hemodialysis therapy with the same mode of dialysis for previous 3 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring hospitalization or interruption of epoetin treatment in previous 6 months;
* significant acute or chronic bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-05-14 (Actual); Primary Completion 2010-06-22 (Actual); Study Completion 2010-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Turkey (Türkiye) (20):
  - Cukurova University Medical Faculty; Internal Medicine, Adana
  - Ankara Research and Training Hospital; The Clinic of Nephrology, Ankara
  - Ankara University School of Medicine; Nephrology, Ankara
  - Faith University School of Medicine; Nephrology, Ankara
  - Hacettepe University Medical Faculty; Department of Internal Medicine, Ankara
  - Baskent University Hospital; Transplantation, Ankara
  - Gazi University School of Medicine; Nephrology, Ankara
  - Adnan Menderes Uni School of Medicine; Physical Therapy & Rehabilitation, Aydin
  - Dicle Uni Medical Faculty; Internal Medicine, Diyarbakır
  - Trakya University Medical Faculty; Internal Medicine; Nephrology, Edirne
  - Firat Uni School Of Medicine; Nephrology, Elâzığ
  - Ataturk University Medical Faculty; Department of Internal Medicine, Erzurum
  - Sisli Etfal Research and Training Hospital; The Clinic of Nephrology, Istanbul
  - Istanbul University Istanbul Medical Faculty; Department of Internal Medicine, Istanbul
  - Marmara Uni School of Medicine; Nephrology, Istanbul
  - Izmir Ataturk Research and Training Hospital; The Clinic of Nephrology, Izmir
  - Dokuz Eylul University School of Medicine; Nephrology, Izmir
  - Erciyes University School of Medicine; Nephrology, Kayseri
  - Inonu Uni School of Medicine, Malatya
  - Mersin University Medical Faculty, Mersin

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 participants were enrolled in this study conducted from 14 May 2008 to 22 June 2010 at 20 centers in Turkey.
Period: Overall Study
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Started | 132
Completed | 102
Not Completed | 30
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 14
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the safety population which included all participants who received at least one dose C.E.R.A. and underwent a safety follow-up, whether withdrawn prematurely or not.
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Their Mean Hemoglobin Concentration Within +/- 1.0 Gram/Deciliter of Their Reference Hemoglobin Concentration and Between 10.0 and 12.0 Gram/Deciliter During the Efficacy Evaluation Period
Description: The reference hemoglobin (Hb) value was taken as the time adjusted average of all Hb assessments during the SVP (Week -4 to Week 0). The time adjusted average Hb concentration of all the values recorded during the efficacy evaluation period (EEP) was calculated for each participant and their reference Hb concentration was subtracted from this value. The percentage of participants maintaining their average Hb concentration during the EEP within +/- 1 gram/deciliter (g/dL) of their reference Hb concentration and between the Hb range 10.0 -12.0 g/dL is presented. The EEP was defined as Week 16 to Week 24. Data missing at the end of the EEP was handled using the last value carried forward method, including any data missing due to withdrawal of participants following red blood cells (RBC) transfusion.
Time Frame: EEP (Week 16 to Week 24)
Population: The per protocol (PP) population included all participants who received at least one dose C.E.R.A. and underwent a safety follow-up except who had < 3 recorded Hb values and had inadequate iron status during EEP, missed C.E.R.A administration during Weeks 16-24, and/or who withdrawn before the end of EEP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- C.E.R.A. 120, 200, or 360 mcg: Eligible participants were administered Continuous Erythropoietin Receptor Activator (C.E.R.A.) at a dose of 120, 200, or 360 microgram (mcg), intravenously (IV), every 4 weeks i.e. Weeks 4, 8, 12, 16 and 20 but not on Weeks 24 and 28 . The initial dose of C.E.R.A.was based on the last dose of the previous Erythropoiesis Stimulating Agent (ESA). The ESA therapy was administered from enrollment to the 4 weeks stability verification period (SVP), weekly, either as epoetin (<8000 IU, 8000-16000 IU, or >16000 IU) or darbepoetin alpha (<40 mcg, 40-80 mcg, or >80 mcg). A telephone follow-up visit took place 4 weeks after the end of C.E.R.A. treatment (Week 28).
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 84
Percentage of participants | 46.43 [35.47 to 57.65]

2. Secondary Outcome: Mean Change in Hemoglobin Concentration Between the Stability Verification Period and the Efficacy Evaluation Period
Description: The mean change in the time-adjusted average Hb concentration between the two study periods The Stability Verification Period (SVP) and EEP is presented. The SVP was defined as Week -4 to Week 0. The EEP was defined as Week 16 to Week 24.
Time Frame: SVP (Week -4 to Week 0) and EEP (Week 16 to Week 24)
Population: The Intention to treat (ITT) population included participants who received at least one dose of C.E.R.A. at Week 0 and for whom data for at least one follow-up variable (adverse event) was available.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 127
g/dL | 0.29 (1.08)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within the Range of 10.0-12.0 Gram/Deciliter Throughout the Efficacy Evaluation Period
Description: The time adjusted average Hb concentration of all the values recorded during the EEP was calculated for each participant. The percentage of participants maintaining their average Hb concentration during the EEP within the Hb concentration range of 10.0-12.0 g/dL is presented. The EEP was defined as Week 16 to Week 24.
Time Frame: EEP (Week 16 to Week 24)
Population: The ITT population included participants who received at least one dose of C.E.R.A. at Week 0 and for whom data for at least one follow-up variable was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 127
Percentage of participants | 51.18 [42.16 to 60.15]

4. Secondary Outcome: Median Time Spent in the Hemoglobin Range 10.0-12.0 Gram/Deciliter During the Efficacy Evaluation Period
Description: The Hb concentration was recorded for all the participants during the EEP. The median time spent (in days) by participants in the target range (10.0-12.0 g/dL) during the EEP is presented. The EEP was defined as Week 16 to Week 24.
Time Frame: EEP (Week 16 to Week 24)
Population: The ITT population included participants who received at least one dose of C.E.R.A. at Week 0 and for whom data for at least one follow-up variable was available. Participants with available data at the time of assessment were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 104
days | 38.0 [21.5 to 51]

5. Secondary Outcome: Mean C.E.R.A. Dose Required to Maintain Hemoglobin Level Within the Range 10.0-12.0 Gram/Deciliter Throughout the Efficacy Evaluation Period
Description: The mean dose of C.E.R.A. required to maintain Hb level between 10.0-12.0 g/dL during the EEP was calculated per participant and then summarized. The EEP was defined as Week 16 to Week 24. However, C.E.R.A. was not administered at the Week 24 visit. Therefore, the time period for calculation of mean C.E.R.A. dose during EEP is from Week 16 to Week 20.
Time Frame: EEP (Week 16 to Week 20)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 33
mcg | 103.5 (46.95)

6. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustments in C.E.R.A. During the Dose Titration Period and Efficacy Evaluation Period
Description: Dose adjustments were necessary when Hb increased or decreased by a clinically significant amount. The dose of C.E.R.A. was adjusted to maintain the individual participant's Hb within a range of +/- 1.0 g/dL of the reference Hb concentration and between 10.0 and 12.0 g/dL throughout the dose titration period (DTP) and the EEP (Week 1 to Week 24). The reference Hb value was taken as the time adjusted average of all Hb assessments during the SVP (Week -4 to Week 0).
Time Frame: DTP (Week 1 to Week 16), EEP (Week 16 to Week 24)
Population: The ITT population included participants who received at least one dose of C.E.R.A. at Week 0 and for whom data for at least one follow-up variable was available. Participants with available data at the time of assessment were included in the analysis. n = number of participants with available data at the time of assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 127
Percentage of participants
  DTP, n = 127 | 75.6
  EEP, n = 107 | 36.4

7. Secondary Outcome: Mean Monthly Dose of C.E.R.A. During the Dose Titration Period and Efficacy Evaluation Period
Description: The mean monthly dose of C.E.R.A. administered during the DTP and EEP was calculated per participant and then summarized.
Time Frame: DTP (Week 1 to Week 16), EEP (Week 16 to Week 24)
Population: The ITT population included participants who received at least 1 dose of C.E.R.A. at Week 0 and for whom data for at least one follow-up variable was available. Participants with available data at the time of assessment were included in the analysis. n = number of participants with available data at the time of assessment.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 127
mcg
  During DTP, n = 127 | 121.6 (47.13)
  During EEP, n = 107 | 112.4 (76.78)

8. Secondary Outcome: Mean Change From Baseline in Erythrocyte Mean Corpuscular Volume at Week 16 and Week 24
Description: Mean change from Baseline in erythrocyte mean corpuscular volume (MCV) was calculated as the value at a specific week during the study minus the BL value. The Baseline was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: The safety population included all participants who received at least one dose of C.E.R.A. and underwent a safety follow-up, whether withdrawn prematurely or not. Participants with available data at the time of assessment were included in the analysis. n = number of participants with available data at the time of assessment.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 102
Femtoliter
  Change from BL to Week 16, n = 102 | -2.02 (3.58)
  Change from BL to Week 24, n = 95 | -1.26 (3.77)

9. Secondary Outcome: Mean Change From Baseline in Hematocrit at Week 16 and Week 24
Description: The hematocrit, also called packed cell volume or erythrocyte volume fraction, is the volume percentage of red blood cells in the blood. Mean change from Baseline (BL) in hematocrit was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 104
percentage of red blood cells
  Change from BL to Week 16, n = 104 | 0.00 (0.04)
  Change from BL to Week 24, n = 99 | 0.01 (0.03)

10. Secondary Outcome: Mean Change From Baseline in Hemoglobin at Week 16 and Week 24
Description: Mean change from BL in hemoglobin was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 104
g/dL
  Change from BL to Week 16, n = 104 | -0.00 (1.16)
  Change from BL to Week 24, n = 98 | 0.22 (1.04)

11. Secondary Outcome: Mean Change From Baseline in Leucocytes and Platelet at Week 16 and Week 24
Description: Mean change from BL in for each parameter (leucocytes and platelet) was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of cells x 10^9/L
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 102
Number of cells x 10^9/L
  Leucocytes, Change from BL to Week 16, n = 102 | 0.27 (2.21)
  Leucocytes, Change from BL to Week 24, n = 95 | -0.03 (1.58)
  Platelet, Change from BL to Week 16, n = 102 | 2.56 (51.21)
  Platelet, Change from BL to Week 24, n = 96 | 0.17 (55.01)

12. Secondary Outcome: Mean Change From Baseline in Ferritin at Week 16 and Week 24
Description: Mean change from BL in ferritin was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: microgram/liter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 93
microgram/liter
  Change from BL to Week 16, n = 93 | 20.80 (283.54)
  Change from BL to Week 24, n = 75 | 31.51 (385.22)

13. Secondary Outcome: Mean Change From Baseline in Iron, Total Iron Binding Capacity, and Creatinine at Week 16 and Week 24
Description: Mean change from BL in each parameter [iron, total iron binding capacity (TIBC), and creatinine] was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 98
micromole/Liter
  Iron, Change from BL to Week 16, n = 98 | 2.08 (6.87)
  Iron, Change from BL to Week 24, n = 93 | 1.15 (6.07)
  TIBC, Change from BL to Week 16, n = 84 | 0.24 (7.09)
  TIBC, Change from BL to Week 24, n = 80 | 0.05 (8.25)
  Creatinine, Change from BL to Week 16, n = 2 | -20.33 (363.80)
  Creatinine, Change from BL to Week 24, n = 92 | 16.73 (218.73)

14. Secondary Outcome: Mean Change From Baseline in Transferrin and Albumin at Week 16 and Week 24
Description: Mean change from BL in each parameter (transferrin and albumin) was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram/liter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 98
gram/liter
  Transferrin, Change from BL to Week 16, n = 33 | 0.19 (0.46)
  Transferrin, Change from BL to Week 24, n = 29 | 0.09 (0.32)
  Albumin, Change from BL to Week 16, n = 98 | 0.13 (3.92)
  Albumin, Change from BL to Week 24, n = 93 | -0.22 (4.58)

15. Secondary Outcome: Mean Change From Baseline in Transferrin Saturation at Week 16 and Week 24
Description: Mean change from BL in transferrin saturation (TSAT) was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of TSAT
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 89
Percentage of TSAT
  Change from BL to Week 16, n = 89 | 4.11 (20.35)
  Change from BL to Week 24, n = 86 | 2.41 (20.18)

16. Secondary Outcome: Mean Change From Baseline in C-Reactive Protein at Week 16 and Week 24
Description: Mean change from BL in C-reactive protein was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 88
milligram/liter
  Change from BL to Week 16, n = 88 | 1.92 (20.64)
  Change from BL to Week 16, n = 81 | -1.43 (20.71)

17. Secondary Outcome: Mean Change From Baseline in Phosphate and Potassium at Week 16 and Week 24
Description: Mean change from BL in each parameter (phosphate and potassium) was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimole/liter
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 97
millimole/liter
  Phosphate, Change from BL to Week 16, n = 97 | 0.04 (0.54)
  Phosphate, Change from BL to Week 24, n = 94 | 0.06 (0.62)
  Potassium, Change from BL to Week 16, n = 94 | -0.04 (0.93)
  Potassium, Change from BL to Week 24, n = 95 | -0.02 (0.93)

18. Secondary Outcome: Mean Change From Baseline in Weight at Week 16 and Week 24
Description: Mean change from BL in weight was calculated as the value at a specific week during the study minus the BL value. The BL was defined as Week -4 to Week 0.
Time Frame: BL (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 103
kilogram
  Change from BL to Week 16, n = 103 | 0.5 (4.17)
  Change from BL to Week 24, n = 100 | 0.7 (4.24)

19. Secondary Outcome: Mean Change in From Baseline in Blood Pressure at Week 16 and Week 24
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured before blood sampling and C.E.R.A. administration. Blood pressure was assessed both before and after the dialysis session for participants undergoing hemodialysis. Change from BL in blood pressure was calculated as the value at a specific week (W) during the study minus the BL value. The baseline was defined as Week -4 to Week 0.
Time Frame: Baseline (Week -4 to Week 0), Week 16, and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 105
Millimeters of Mercury
  SBP Before Dialysis,Change from BL to W 16,n = 105 | 2.1 (14.94)
  DBP Before Dialysis,Change from BL to W 16,n = 105 | 2.4 (10.61)
  SBP Before Dialysis,Change from BL to W 24,n = 101 | 3.0 (15.46)
  DBP Before Dialysis,Change from BL to W 24,n = 101 | 2.2 (11.24)
  SBP After Dialysis,Change from BL to W 16, n = 100 | -0.3 (17.54)
  DBP After Dialysis,Change from BL to W 16, n = 100 | 1.7 (10.91)
  SBP After Dialysis,Change from BL to W 24, n = 95 | 1.0 (15.88)
  DBP After Dialysis, Change from BL to W 24, n = 95 | 1.8 (10.94)

20. Secondary Outcome: Number of Participants Taking Concomitant Medications
Description: The number of participants taking different classes of concomitant medications at any time following enrollment into the study is presented.
Time Frame: Up to Week 28
Population: The safety population included all participants who received at least one dose of C.E.R.A. and underwent a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 131
Number of participants
  Antibacterials for systemic use | 13
  Vitamins | 13
  Vaccines | 7
  Agents acting on the renin-angiotensin system | 5
  Analgesics | 4
  Antianemic preparations | 4
  Antithrombotic agents | 4
  Drug for acid related disorders | 4
  Mineral supplements | 4
  Other | 4

21. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 28
Population: as for outcome 20
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 131
Number of participants
  Number of participants with any AE | 44
  Number of participants with any SAE | 13

22. Secondary Outcome: Number of Participants With Reports of Anti-erythropoietin Antibodies
Description: The number of participants with Anti-epoetin antibodies is presented.
Time Frame: Up to Week 24
Population: as for outcome 20
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 131
Number of participants | 0

23. Secondary Outcome: Number of Participants Who Received Red Blood Cell Transfusions During the Dose Titration Period and Efficacy Evaluation Period
Description: Red blood cell transfusions were permitted during the DTP and EEP (Week 1 to Week 24) in case of medical need. All participants requiring a blood transfusion were withdrawn from the study. The number of participants who were administered RBC transfusions during the DTP and EEP is presented.
Time Frame: Week 1 to Week 24
Population: as for outcome 20
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Number analyzed (Participants) | 131
Number of participants
  During DTP | 1
  During EEP | 0

ADVERSE EVENTS:
Time Frame: Up to Week 28
Description: Adverse events were analyzed for the safety population which included all participants who received at least one dose of C.E.R.A. and underwent a safety follow-up, whether withdrawn prematurely or not.
Arm/Group | C.E.R.A. 120, 200, or 360 mcg
Serious Adverse Events (participants affected / at risk) | 13/131
Other Adverse Events (participants affected / at risk) | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. 120, 200, or 360 mcg (N=131)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal transplant (Surgical and medical procedures) | 1
Subclavian vein thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Low number of participants completed the study as per the protocol. Administration of iron (oral/IV) was as per discretion of individual centers; therefore, C.E.R.A. responses have been limited by iron levels too low for efficient erythropoiesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.